CLINICAL TRIAL: NCT00484107
Title: A Postmarketing Surveillance Study Evaluating the Tolerability and Safety of PREMARIN VAGINAL CREAM in Indian Postmenopausal Women
Brief Title: Tolerability & Safety of Premarin Vaginal Cream in Indian Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0713V-101833
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Postmenopause
MeSH Terms: interventions — Estrogens, Conjugated (USP)

INTERVENTIONS:
Drug: Conjugated Estrogen Cream (Premarin®)

SUMMARY:
This post-marketing study will provide local safety and tolerance data on the use of Premarin® vaginal cream.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom Premarin vaginal cream is indicated.
* In the opinion of the investigator, sufficient intelligence and motivation for the patient to continue throughout the study.
* Provide signed informed consent.

Exclusion Criteria:

* Patients not willing to give informed consent.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-09; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer